CLINICAL TRIAL: NCT02630537
Title: Clinical Validation of Lophius Kits T-Track® CMV and T-Track® EBV to Assess the Functionality of Cell-mediated Immunity (CMI) in Hemodialysis Patients
Brief Title: Validation of Lophius Kits T-Track® CMV and T-Track® EBV in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Lophius Biosciences GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: LB-A1 (UREA-CMV-EBV)
Record Dates: First submitted 2015-12-07; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Renal Failure Chronic Requiring Dialysis
Keywords: Cytomegalovirus; Epstein- Barr virus; Cell-mediated immunity; T-Track® CMV; T-Track® EBV; hemodialysis; ELISpot
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Cell-mediated immunity (CMI) and in particular T cells play a critical role in the rejection of transplanted organs. Thus, in transplant recipients a life-long and individualized immunosuppressive medication is required to avoid graft rejection. However, a too weak suppression of CMI causes acute and chronic graft damage leading to transplant loss, whereas a too potent suppression of CMI supports opportunistic infections and reactivation of persistent viruses.

One of the biggest challenges in the field of transplantation is to provide a personalized immunosuppressive and antiviral therapy based on reliable assessment and monitoring of CMI. This could lead to a reduction of graft rejections and virus reactivations in transplant recipients.

With the development of both assays T-Track® CMV and T-Track® EBV, Lophius Biosciences GmbH has implemented its novel proprietary T-activation technology for an improved assessment of the functionality of CMI in cytomegalovirus (CMV)- and/or Epstein-Barr virus (EBV)-seropositive individuals. In contrast to other existing systems the Lophius assays open up the opportunity to characterize the functionality of CMI as an entire network.

The planned clinical multicenter study aims to verify the suitability of the two assays for a reliable assessment of the functionality of CMI.

Hemodialysis patients have been identified as an appropriate patient cohort for investigating the clinical sensitivity of the Lophius assays as these patients closely resemble kidney transplant recipients prior to an immunosuppressive therapy.

The determination of the functional CMI in the course of an immunosuppressive treatment may in future enable physicians to optimize the individual immunosuppressive and antiviral therapy in transplant recipients to reduce the risk of rejection as well as virus reactivations and associated diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patient being hemodialysis-dependent due to end-stage kidney disease
* Male or female patient at least 18 years of age
* Written informed consent

Exclusion Criteria:

* Patient requires ongoing dosing with a systemic immunosuppressive drug
* Patient has received immunosuppressive therapy within the last three month
* Patient is known to be positive for HIV or suffering from chronic hepatitis infections
* Patient has significant uncontrolled concomitant infections or other unstable medical conditions that could interfere with the study objectives
* Patient has any form of substance abuse, psychiatric disorder or condition that, in the opinion of the investigator may invalidate communication with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient being hemodialysis-dependent due to end-stage kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percentage of CMV or EBV seropositive hemodialysis patients showing significant numbers of functional CMV or EBV-protein-reactive blood leucocytes applying T-Track® CMV or T-Track® EBV | 1 day
  Determination of the clinical sensitivity of T-Track® CMV and T-Track® EBV. T-Track® assays are based on the stimulation of peripheral blood mononuclear cells (PBMC) with preselected immunodominant T-activated proteins derived from the human Cytomegalovirus (CMV) and the Epstein-Barr-Virus (EBV) and the subsequent quantification of IFN-gamma producing blood leucocytes (Lophius biomarker for assessing the functionality of CMI) applying ELISpot technology.

SECONDARY OUTCOMES:
Percentage of CMV or EBV seropositive hemodialysis patients showing significant numbers of functional CMV or EBV-protein-reactive blood leucocytes applying EBV and CMV peptide-loaded Pro5® Pentamers and the Quantiferon® CMV assay | 1 day
  The comparison of the suitability of T-Track® CMV and T-Track® EBV to EBV and CMV peptide-loaded Pro5® Pentamers and the Quantiferon® CMV assay (commercially available competing products)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Banas, Prof., Principal Investigator — University Medical Center Regensburg

REFERENCES:
- [Derived] Banas B, Boger CA, Luckhoff G, Kruger B, Barabas S, Batzilla J, Schemmerer M, Kostler J, Bendfeldt H, Rascle A, Wagner R, Deml L, Leicht J, Kramer BK. Validation of T-Track(R) CMV to assess the functionality of cytomegalovirus-reactive cell-mediated immunity in hemodialysis patients. BMC Immunol. 2017 Mar 7;18(1):15. doi: 10.1186/s12865-017-0194-z. PMID 28270092